CLINICAL TRIAL: NCT07344051
Title: A Randomized, Double-Blind, Placebo-Controlled Phase II Clinical Trial Evaluating the Efficacy and Safety of QLS12010 Capsules in Adult Participants With Moderate-to-Severe Atopic Dermatitis
Brief Title: A Phase II Study of QLS12010 Capsules in Adults With Moderate to Severe Atopic Dermatitis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QLS12010-201
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Moderate-to-severe Atopic Dermatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- QLS12010 Capsule Dose 1 Group (Experimental)
  Interventions: Drug: QLS12010
- QLS12010 Capsule Dose 2 Group (Experimental)
  Interventions: Drug: QLS12010
- QLS12010 Capsule Dose 3 Group (Experimental)
  Interventions: Drug: QLS12010
- Placebo Group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QLS12010 — QLS12010 oral capsule
  Arms: QLS12010 Capsule Dose 1 Group; QLS12010 Capsule Dose 2 Group; QLS12010 Capsule Dose 3 Group
Drug: Placebo — Matching placebo oral capsule
  Arms: Placebo Group

SUMMARY:
This trial was designed to evaluate the efficacy and safety of QLS12010 Capsules in adults with moderate-to-severe atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

1. At screening, the diagnosis of atopic dermatitis (AD) shall meet the Hanifin-Rajka criteria, with a duration of AD ≥ 1 year prior to baseline;
2. At screening and baseline: Eczema Area and Severity Index (EASI) score ≥ 16 points, Investigator's Global Assessment (IGA) score ≥ 3 points, and body surface area (BSA) affected by AD ≥ 10%;
3. At baseline: Weekly mean score of Pruritus Numerical Rating Scale (PP NRS) ≥ 4 points (with daily PP NRS scores recorded on at least 4 days within the 1 week prior to baseline);

Exclusion Criteria:

1. Participants with other medical conditions (excluding AD) that, as determined by the investigator, may interfere with the evaluation of efficacy or safety in this study, including but not limited to psoriasis, seborrheic dermatitis, systemic lupus erythematosus, moderate-to-severe acne, infectious folliculitis, etc.;
2. History of severe cardiovascular and cerebrovascular diseases occurring within 6 months prior to screening, including but not limited to unstable angina pectoris, New York Heart Association (NYHA) Class III or IV heart failure, myocardial infarction, cardiomyopathy, cerebral hemorrhage, acute cerebral infarction, etc.;
3. Participants with a history of prior use of IRAK4 degraders, small-molecule IRAK4 inhibitors, or similar agents;
4. Participants who have received treatment with other investigational products (IPs) within 3 months or 5 half-lives (whichever is longer) prior to screening;
5. Pregnant or lactating women, or participants with a positive pregnancy test result at screening;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-04-05 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Percentage Change in Eczema Area and Severity Index (EASI) Score from Baseline at Week 16. | At Week 16.
  The minimum EASI score is 0, and the maximum EASI score is 72. A score of 0 indicates clear or no eczema; a greater score indicates more severe disease.